CLINICAL TRIAL: NCT06246097
Title: INVESTIGATION of EXPRESSION of C-TERMINAL CROSS-LINKING TELOPEPTIDE of TYPE I COLLAGEN(CTXI) LEVELS IN SALIVA WITH EARLY and DELAYED LOADING of DENTAL IMPLANTS
Brief Title: INVESTIGATION of EXPRESSION of CTXI LEVELS IN SALIVA WITH EARLY and DELAYED LOADING of DENTAL IMPLANTS
Status: Completed | Type: Observational
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Dania Hamid, Dr. Dania Hamid, Dow University of Health Sciences
Other Study IDs: dowuhs123
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Dental Implant, Periotest, CTX,Delayed Loading, ELISA, Early Loading, Saliva

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: early loading of dental implants within a month
- group 2: delayed loading of dental implants within 3 months

SUMMARY:
Background:

Implants are commonly used as a treatment choice for partially dentate or in edentulous patients. Currently, no specific biomarker to assess the bone status around the dental implants of healthy patients has been reported to further evaluate bone deposition, resorption and stability. CTX (C-terminal telopeptide) is a known specific biomarker for bone resorption. CTX levels evaluation in serum and urine of patients with bisphosphonates treatment has already been reported. However, its levels in saliva of healthy patients with dental implants has not been investigated, so far.

Objectives:

The aim of this study is to evaluate salivary CTX levels in dental implants with early and delayed loading and to compare it with the values of mechanical stability test (Periotest).

Methods:

Patients coming to OPD of Oral Surgery department of Dow International Dental College (DIDC) and are willing for placement of implant in the posterior molar area of mandible will be enrolled in the study. Informed consent will be taken from each patient for participation in the study. Dental implants placement will be performed according to the standard protocols. All patients will be assessed for implant stability on the day of surgery, at 1 month, 2 month and 3 months by Periotest assessment. Also, saliva will be collected and stored from same patients. Later, ELISA will be performed for expressional analysis of CTX.

DETAILED DESCRIPTION:
40 Patients coming to OPD of Dow International Dental College for implant placement in posterior mandible (molar area) will be recruited in the study.

Dental implants available in the Outpatient Department (OPD) of Dow International Dental College (DIDC) will be placed in patients. Dental implants will be placed according to the standard protocols by Dr. Shaheen Ahmed.

Patients will be divided in two groups. Group A patients will be early loaded, and group B will be conventional loaded with prosthesis.

Each patient will be evaluated for implant stability after the surgery, at 1 month, 2 months and 3 months with the help of Periotest.

Saliva will be collected from patients in both the groups before placement of implant and on the same days as of Periotest evaluations after surgery. Saliva will be processed and immediately stored at -80oC. Later sandwich ELISA will be performed for expressional analysis of CTX.

Levels of CTX before implant surgery will be served as reference value in this study.

2.9.1 Saliva Collection Method:

Whole unstimulated saliva (WUS) will be collected from both the study groups. The process of saliva collection is as follows:

* Salivary samples will be collected between 9-11 am to minimize diurnal variations in salivary flow and changes in the sialo chemistry.
* Patients will be asked to refrain from smoking, drinking and chewing at least one hour before saliva collection to avoid interference of water and food with the analysis.
* To remove any food debris from mouth, the patients will be asked to wash the mouth with water before saliva collection.
* After rinsing thoroughly, an interval of at least 10 minutes will be given before the collection of saliva samples to avoid sample dilution.
* Patients will be asked to spit the saliva in a sterilized falcon tube of 15mL.
* Approximately 2-5 mL of saliva will be collected from each patient.
* Patient will be informed and told not to cough up mucus.
* After saliva collection, samples will be immediately taken to the laboratory for further processing.
* Salivary samples will be centrifuged at 8000rpm for 15 min at 4˚C to remove any cell debris and supernatant will be collected.
* The collected supernatant will be aliquoted into microtubes of 1ml and will be stored at -80°C until further analysis (processing time of saliva will be kept lowest as possible).

2.9.2 Salivary Analysis:

Enzyme Linked Immunosorbent Assay (Sandwich Technique):

CTX levels in salivary samples of all the groups will be analyzed by sandwich ELISA (Enzyme Linked Immunosorbent Assay) technique. ELISA testing will be performed by using CTX kit according to manufacturer's instruction. The plate pre-coated with antibody specific to Human CTX will be provided with the kit. Standards or samples are added to the micro ELISA plate wells which allows CTX to bind to its specific antibody. After removing unbound sample, biotinylated CTX detection antibody will be added followed by washing with the buffer. After washing, plate will be incubated with Streptavidin-Horseradish Peroxidase (HRP) that will binds to detection antibody. After incubation, unbound Streptavidin-HRP will be washed away. Finally, substrate solution will be added. The intensity of color developed is proportional to the amount of human CTX present in the sample. The reaction will be stopped by the addition of stop solution and absorbance will be measured spectrophotometrically at 450 nm wavelength. The concentration of CTX in samples is obtained by comparing absorbance of samples to the standards.

ELISA will be performed by principal investigator of the study with the help of her Co-supervisor in DRIBBS (Dow Research Institute of Biotechnology and Biomedical Sciences).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects of age 18 and above.
* Patients who have consented to be part of the study.
* Patients in whom only posterior mandibular implants are to be placed.

Exclusion Criteria:

* • Patients with known bone diseases such as osteoarthritis, osteoporosis etc.

  * Patient with uncontrolled diabetes and uncontrolled hypertension etc.
  * Patients who need maxillary implants.
  * Patients treated with oral cancer.
  * Patients who are given implants in fresh extraction sockets.
  * Patients in whom bone augmentation is needed.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients coming to OPD of Dow International Dental College for implant placement in posterior mandible (molar area) will be recruited in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
c terminal telopeptide of type I collagen | 3 monts
  bone resorption biomarker

CONTACTS AND LOCATIONS:
Locations (1):
- Dania Hamid, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Elani HW, Starr JR, Da Silva JD, Gallucci GO. Trends in Dental Implant Use in the U.S., 1999-2016, and Projections to 2026. J Dent Res. 2018 Dec;97(13):1424-1430. doi: 10.1177/0022034518792567. Epub 2018 Aug 3. PMID 30075090
- [Background] Guglielmotti MB, Olmedo DG, Cabrini RL. Research on implants and osseointegration. Periodontol 2000. 2019 Feb;79(1):178-189. doi: 10.1111/prd.12254. PMID 30892769
- [Background] Esposito M, Siormpas K, Mitsias M, Bechara S, Trullenque-Eriksson A, Pistilli R. Immediate, early (6 weeks) and delayed loading (3 months) of single implants: 4-month post-loading from a multicenter pragmatic randomised controlled trial. Eur J Oral Implantol. 2016;9(3):249-260. PMID 27722223
- [Background] Zhu Y, Zheng X, Zeng G, Xu Y, Qu X, Zhu M, Lu E. Clinical efficacy of early loading versus conventional loading of dental implants. Sci Rep. 2015 Nov 6;5:15995. doi: 10.1038/srep15995. PMID 26542097
- [Background] Le Guehennec L, Soueidan A, Layrolle P, Amouriq Y. Surface treatments of titanium dental implants for rapid osseointegration. Dent Mater. 2007 Jul;23(7):844-54. doi: 10.1016/j.dental.2006.06.025. Epub 2006 Aug 14. PMID 16904738
- [Derived] Hamid D, Ahmed S, Shaikh AH, Nisar S, Memon R, Malik S. Investigation of the expression of the C-terminal cross-linking telopeptide of type I collagen (CTXI) in saliva during early and delayed loading of dental implants. BMC Oral Health. 2025 Jul 2;25(1):1013. doi: 10.1186/s12903-025-05529-x. PMID 40604796